CLINICAL TRIAL: NCT01129973
Title: Profile of Marketing Professional Audiologist Who Works in the Area of Audiology Clinic
Acronym: Audiologist
Status: Completed | Type: Observational
Sponsor: Fortaleza University (Other)
Responsible Party: Marilia Fontenele e Silvia Câmara, University of Fortaleza
Other Study IDs: CLEICE01
Record Dates: First submitted 2010-05-24; First posted 2010-05-25 (Estimated); Last update posted 2010-05-25 (Estimated); Status verified 2010-01

CONDITIONS: Audiologist; Fortaleza
Keywords: speech and language; phonoaudiology; marketing
MeSH Terms: conditions — Speech; Language

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: None Retained — no biospecimens are to be retained.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
the audiology has achieved a great advance, where currently speech pathologists act in private clinics and in public services, in addition to schools, colleges and universities. To observe the development of the area of Audiology in Brazil, we note that there is a growing number of new audiology procedures. In 1980 the practice of audiology was limited in hospitals, offices and private clinics, and in 1988 due to a new constitution that devoted attention to protection of health of workers, opened-if more than one field of work, the audiology occupational, because of the hearing losses induced by noise

DETAILED DESCRIPTION:
The area of audiology referred-if the science of hearing, auditory processing and corporal balance. The speech pathologist, Especialista em Audiologia, identifies, assesses and rehabilitation, empowering people with disabilities peripheral or central auditory, influencing the emergence of human communication disorders, as well as the balance disorders

ELIGIBILITY:
Inclusion Criteria:

* the professionals working with clinical audiology

Exclusion Criteria:

* the professionals who do not act in the city of Fortaleza or refuse to sign the Term of Free and Informed Consent

Ages: 24 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: replied to the questionnaire speech pathologists, of both sexes, active in the area of audiology clinic, of the city of Fortaleza, Ceará.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2010-01; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cleiciane M Braga, Graduate, Principal Investigator — Fortaleza University